CLINICAL TRIAL: NCT06498583
Title: Effect of Ultrasound-guided Erector Spinae Plane Block on Postoperative Pain and Sleep Quality of Infants With Congenital Pulmonary Cystic Disease After Thoracoscopic Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Lei Xiaoming (Other)
Responsible Party: Sponsor-Investigator, Lei Xiaoming, chief physician, Xibei Hospital
Organization: Xibei Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2024-015
Record Dates: First submitted 2024-06-28; First posted 2024-07-12 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Cystic Adenomatoid Malformation of Lung, Congenital; Bronchopulmonary Sequestration; Bronchogenic Cyst
MeSH Terms: conditions — Cystic Adenomatoid Malformation of Lung, Congenital; Bronchopulmonary Sequestration; Bronchogenic Cyst | interventions — Ropivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- E group (Experimental)
  Interventions: Drug: Ropivacaine; Procedure: erector spinae plane block
- P group (Experimental)
  Interventions: Drug: Ropivacaine; Procedure: Incision infiltration of local anesthesia

INTERVENTIONS:
Drug: Ropivacaine — 0.25 % ropivacaine ( 0.5ml / kg )
Procedure: erector spinae plane block — After the operation, unilateral erector spinae plane block was performed at the T5 level under ultrasound guidance.
  Arms: E group
Procedure: Incision infiltration of local anesthesia — After the operation, Incision infiltration of local anesthesia is performed around the surgical incisions.
  Arms: P group

SUMMARY:
This study intends to evaluate the effect of erector spinae plane block on postoperative analgesia and sleep quality in infants with congenital cystic pulmonary disease after thoracoscopic surgery, and provides reference for perioperative pain treatment in children.

DETAILED DESCRIPTION:
Severe pain may occur after pediatric thoracic surgery, such as skin incision, rib traction, drainage tube placement, or intercostal nerve dysfunction caused by suture. Pain may cause weakened coughing power to clear secretions, decreased functional residual capacity, leading to pulmonary complications such as atelectasis and pneumonia, and postoperative acute pain develops into chronic pain. It has been reported that postoperative sleep disorders are associated with increased pain scores, which are very unfavorable for postoperative rehabilitation of pediatric patients. In clinical practice, because infants cannot accurately describe pain, their postoperative pain management may not be sufficient and has not received enough attention. But, some studies have shown that infants may feel more severe pain than adults, and the pain has a more obvious and lasting effect on infants and young children than on adults.

Congenital pulmonary cystic disease is a rare congenital pulmonary developmental abnormality in clinic. It can't heal itself and is easy to cause various complications. Once diagnosed, surgical treatment should be considered immediately.

In the past experience, thoracic epidural block and thoracic paravertebral nerve block are commonly used for postoperative analgesia in thoracic surgery, but they have taboos such as abnormal coagulation function, high technical requirements and potential risks of serious complications.

Since the erector spinae plane block (ESPB) was first reported and successfully implemented in 2016, because it is far away from the neural axis, major vascular structures, pleura and other structures, with a lower possibility of complications, simpler operation and higher safety, it has been widely used in perioperative analgesia and acute and chronic pain in cardiothoracic surgery, breast surgery, abdominal surgery, spinal surgery, etc. However, the reports on pediatric patients are still mainly case reports, and there is a lack of large-sample randomized controlled clinical trials. Therefore, this study intends to perform erector spinae plane block under ultrasound guidance to observe the effect on postoperative analgesia and sleep quality in pediatric thoracoscopic surgery.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) status I-II
* age 1 month - 12 mouths old
* preoperative diagnosis was congenital cystic lung disease
* thoracoscopic lung lesion resection(lung lobectomy or segmentectomy)

Exclusion Criteria:

* patient with a history of allergy to amide local anesthetics
* family members refused to participate in the study.
* combined congenital heart disease
* patient with skin damage or infection at the proposed puncture site
* patients with scoliosis

Ages: 1 Month to 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2024-09-05 (Estimated); Primary Completion 2025-02 (Estimated); Study Completion 2025-02 (Estimated)

PRIMARY OUTCOMES:
postoperative FLACC score | 2, 4, 6, 12, 24, 48 hours after operation

SECONDARY OUTCOMES:
Postoperative sleep quality score | 1, 2, 3, 4, 5, 6, 7 days after operation
  The Pittsburgh Sleep Quality Index was used to evaluate the sleep quality of children 7 days after surgery.
Number of participants with emergence agitation as assessed by PAED | from extubation to the child is sent back to the ward, an average of 40 minutes
  The Pediatric Anesthesia Emergence Delirium (PAED) was used to evaluate emergence agitation after extubation in post-anesthesia care unit.
the amount of postoperative rescue analgesia ( with a FLACC score of >4) | 2, 4, 6, 12, 24, 48 hours after operation
  ibuprofen (5-10mg/kg) was intravenously administered as rescue analgesia.

CONTACTS AND LOCATIONS:
Overall Officials: Xiaoming Lei, chief physician, Study Chair — Second Affiliated Hospital of Xi 'an Jiaotong University
Locations (1):
- Second Affiliated Hospital of Xi 'an Jiaotong University, Xi’an, Shanxi, China